CLINICAL TRIAL: NCT00688857
Title: A Randomized, Open-label, Multi-dose Crossover Study Assessing the Pharmacokinetic Profiles of Diazoxide Choline Coated Versus Uncoated Formulations in Healthy Volunteers
Brief Title: Open-label Pharmacokinetic Study of Diazoxide Choline Coated vs. Uncoated Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Essentialis, Inc. (Industry)
Collaborators: Cetero Research, San Antonio (Network)
Responsible Party: Neil M Cowen, PhD/Chief Scientific Officer, Essentialis, Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PK008
Record Dates: First submitted 2008-05-28; First posted 2008-06-03 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-11

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Diazoxide choline controlled-release coated tablets administered orally once daily (Days 1 through 8). Diazoxide choline controlled-release uncoated tablets administered orally once daily (Days 9 through 16).
  Interventions: Drug: Diazoxide choline
- B (Experimental): Diazoxide choline controlled-release uncoated tablets administered orally once daily (Days 1 through 8). Diazoxide choline controlled-release coated tablets administered orally once daily (Days 9 through 16)
  Interventions: Drug: Diazoxide choline

INTERVENTIONS:
Drug: Diazoxide choline — Diazoxide choline controlled-release coated tablets versus Diazoxide choline controlled-release uncoated tablets administered orally once daily
  Arms: A
Drug: Diazoxide choline — Diazoxide choline controlled-release uncoated tablets versus Diazoxide choline controlled-release coated tablets administered orally once daily
  Arms: B

SUMMARY:
This is a single-center, randomized, open-label, multi-dose crossover study assessing the pharmacokinetic profiles of diazoxide choline coated versus uncoated formulations in healthy volunteers. The primary objective is to compare the pharmacokinetic (PK) profiles of diazoxide choline controlled-release coated tablets versus uncoated tablets in healthy volunteers under fed conditions. Secondary objectives are to assess diazoxide choline pharmacokinetic (PK) parameters under fasted conditions, and to assess the safety and tolerability of diazoxide choline controlled-release coated tablets versus uncoated tablets in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Healthy male and female subjects 18 to 75 years of age
* Body mass index (BMI) between 22-35 kg/m2
* Fasting glucose ≤ 125 mg/dL and HbA1C ≤ 6.5.
* Fasting triglyceride ≥100 mg/dL and ≤ 500 mg/dL
* Not pregnant

Exclusion Criteria:

* Significant underlying medical conditions
* Clinical laboratory test values outside the accepted range
* Smokers, tobacco users, or subjects currently using nicotine products
* Substance abuse
* History of allergic response(s) to diazoxide or related drugs
* Recent significant weight loss
* Use of medication affecting body weight, lipid or glucose metabolism
* Unable to comply with study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Compare the pharmacokinetic (PK) profiles of diazoxide choline controlled-release coated tablets versus uncoated tablets in healthy volunteers under fed conditions. | 16 days

SECONDARY OUTCOMES:
Assess diazoxide choline pharmacokinetic (PK) parameters under fasted conditions | Study days 8 and 16
Assess the safety and tolerability of diazoxide choline controlled-release coated tablets versus uncoated tablets in healthy volunteers. | Entire study

CONTACTS AND LOCATIONS:
Overall Officials: Alan K. Copa, Pharm. D., Principal Investigator — PRACS Institute, Ltd. - Cetero Research
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States